CLINICAL TRIAL: NCT03618277
Title: Identification of Biological Markers and Biometrological Characterization of Melasma
Brief Title: Identification of Biomarkers and Characterization of Melasma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: business strategy
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MELASMAPHYSIOBIOMETRO
Record Dates: First submitted 2018-07-26; First posted 2018-08-07 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2018-08

CONDITIONS: Chloasma
MeSH Terms: conditions — Melanosis | interventions — Biopsy; Photography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intra individual (Other): Before and after being treated by a product (outside the study)
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Micro-biopsies will be performed using a punch of 1 mm in diameter, by pulling the skin at the time of sampling, after disinfection and anesthesia.
  Other Names: Photography

SUMMARY:
Melasma (also called chloasma and pregnancy mask) is characterized by pigmented lesions darker than their usual complexion on the faces of affected subjects.

The physiopathology of melasma is still poorly understood. To date, the factors that favor the onset of melasma appear to be: genetic predisposing factors, changes in sex hormone levels, and sun exposure.

Vascularization as well as elastosis also appear to be increased in skin with melasma.

The aim of this study is to evaluate the different levels of expression of biomarkers between pigmented melasma lesions and surrounding healthy skin when melasma is highly pigmented but also when it is dormant (ie treated melasma, without UV solicitation in the heart of winter). The goal is to identify and better understand the involvement of different genes and proteins and thus offer more specific ways of care, and therefore effective, for the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged 18 to 60 years old included
* Phototype III to IV included according to Fitzpatrick classification
* Informed consent signature
* Subject accepting micro-biopsies on study areas
* Subject with melasma lesions in the face of moderate to severe intensity defined by clinical rating (Physician Global Assesment Static) allowing the realization of micro-biopsies according to the opinion of the investigator

Exclusion Criteria:

* Subject having planned to stay more than 7 consecutive days in a place with a significant increase in the UV index (ski holidays, travel to the tropics, etc.)
* Subject with pigmented facial lesions other than those related to melasma.
* Subject having already presented cicatrization disorders
* Subject having undergone a physical treatment (radiotherapy ...) on the face, during the last 6 months or planned during the study
* Chemical peel, laser treatment or dermabrasion, performed on the face in the 3 months preceding the inclusion visit,
* Application of medication containing hydroquinone or other depigmenting treatments (retinoids, topical steroids) applied to the face in the 2 months prior to the inclusion visit,
* Applying depigmenting cosmetic products to the face within 4 weeks prior to the inclusion visit

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline at Visite 2 : Biomarkers evaluation of melasma, obtained by microbiopsies | Visit 1 (Baseline) and Visit 2 (Day 150 +/- 30 days)
  The expression levels of the biomarkers (transcriptomic and proteomic) of each zone will be measured and compared.
  Transcriptomic analysis will be performed by biochip. Proteomic analysis will be performed by mass spectroscopy.
Change from baseline at Visite 2 : Photographic evaluation of melasma | Visit 1 (Baseline) and Visit 2 (Day 150 +/- 30 days)
  From photographs, the severity of the lesions will be evaluated.
Change from baseline at Visite 2 : Clinical evaluation of melasma by P.G.A. scales | Visit 1 (Baseline) and Visit 2 (Day 150 +/- 30 days)
  Different intensities of melasma will be evaluated by clinical rating : Physician Global Assessment (PGA) Static (4-point scale) and Dynamic (7-point scale).

CONTACTS AND LOCATIONS:
Overall Officials: Didier COUSTOU, Dr, Principal Investigator

IPD SHARING:
Plan to Share IPD: No